CLINICAL TRIAL: NCT03536546
Title: Improving Outcomes for Emergency Department Patients With Alcohol Problems
Acronym: Project GOAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 16-235
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Results first posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Drinking, Alcohol
Keywords: Veterans Health; Intervention, Brief; Peer
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol; Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Veteran peer research assistants will deliver alcohol brief advice in the ED and will initiate conversations with the participant for at least 6-sessions over 2 months post-ED visit. Strengths-based discussions will include a combination of scripted and open-ended content to best facilitate reductions in drinking and engagement across severity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcohol Peer-Mentor Intervention (Experimental): A Veteran Peer research assistant will have contact with a study participant once in person in the emergency department at enrollment, and up to 6 times after enrollment over the course of 2 months. Participants will receive brief advice from a peer. Brief advice content will be based on strengths-based discussions with participants regarding their drinking and personal goals and preferences. Participants will also receive a resource pamphlet on alcohol and other health issues. Follow-up contact will be made by phone. The content of the follow-up peer intervention will be based on the manual developed by the study team to address strengths-based intervention topics.
  Interventions: Behavioral: Alcohol Peer Mentor Intervention
- Brief Advice (Active Comparator): Participants will receive brief substance use advice from a non-peer research staff member in the emergency department. Brief advice content will mirror standard care practices currently provided in VHA when a patient endorses hazardous drinking behaviors. Participants will also receive a resource pamphlet on alcohol and other health issues.
  Interventions: Behavioral: Brief Advice

INTERVENTIONS:
Behavioral: Alcohol Peer Mentor Intervention — A Veteran Peer research assistant will have contact with a study participant once in person in the emergency department at enrollment, and up to 6 times after enrollment over the course of 2 months. Participants will receive brief advice from a peer. Brief advice content will be based on strengths-based discussions with participants regarding their drinking and personal goals and preferences. Participants will also receive a resource pamphlet on alcohol and other health issues. Follow-up contact will be made by phone. The content of the follow-up peer intervention will be based on the manual developed by the study team to address strengths-based intervention topics.
  Other Names: APM
  Arms: Alcohol Peer-Mentor Intervention
Behavioral: Brief Advice — Participants will receive brief substance use advice from a non-peer research staff member in the emergency department. Brief advice content will mirror standard care practices currently provided in VHA when a patient endorses hazardous drinking behaviors. Participants will also receive a resource pamphlet on alcohol and other health issues.
  Other Names: BA
  Arms: Brief Advice

SUMMARY:
The investigators will conduct a study to examine the impact of an alcohol peer-mentor intervention starting in the emergency department (ED) combined with 6 peer booster sessions to reduce hazardous drinking and facilitate primary/specialty care use compared to enhanced usual care. Approximately 450 Veterans with hazardous drinking behaviors will be randomized to one of these two conditions. Follow-up assessments will occur at 3-, 6-, and 12-month post-randomization.

DETAILED DESCRIPTION:
The objective of the study is to conduct a randomized controlled trial to determine the efficacy of an alcohol peer-mentor intervention starting in the ED, combined with a continuing 6-session program of post-ED strengths-based peer mentorship to facilitate reduction in hazardous drinking, and linkage and engagement in primary and/or specialty alcohol treatment services and mental health care, if needed. Project Methods: The study will screen Veterans Affairs (VA) ED patients for hazardous drinking. Those screening positive and who enroll in the study will be randomized to one of two conditions: 1) Alcohol Peer-Mentor (APM) intervention (n=225), or 2) Brief Advice (BA) comparison condition (n=225). Stratified random assignment to conditions will be by sex and presence of AUD (yes/no) defined as a score of 14 for men and 10 for women on the AUDIT. Randomization will proceed in blocks of 10. All participants will also receive written community resource information. Participants randomized to the APM condition will receive peer support to reduce hazardous drinking, and those who meet alcohol use disorder criteria will be coached by the peer and will assist in a warm handoff linkage to addiction treatment.

ELIGIBILITY:
Inclusion Criteria:

Screening:

* Presenting for care in the Ann Arbor Veterans Health Administration (VHA) ED
* Medically stable
* Able to provide informed consent

Enrollment:

* Have an AUDIT-C score of 4 or more for men and 3 or more for women in the prior 3 months, indicating that they meet criteria for hazardous use (NIAAA 2005; World Health Organization)
* Have a telephone and/or the ability to provide information about individuals who can help contact the participant

Exclusion Criteria:

Screening:

* Do not understand English
* Patients in or having received substance abuse treatment in the past 3-months, per medical record
* Patients in or having received peer services in the past 3-months, per medical record
* Pregnant women
* Patients deemed unable to provide informed consent
* Profound psychotic symptoms and/or cognitive deficits that would prevent patients from understanding the content of the intervention and/or assessments

Enrollment:

* Patients currently active in or having received alcohol or other substance abuse treatment in the past 3-months, per self-report screening.
* Patients currently active in or having received peer services in the past 3-months, per self-report screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul N Pfeiffer, MD MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alcohol Peer-Mentor Intervention | Brief Advice
Started | 104 | 101
Completed | 90 | 92
Not Completed | 14 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol Peer-Mentor Intervention | Brief Advice | Total
Number analyzed (Participants) | 104 | 101 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (15.7) | 53.9 (16.8) | 53.7 (16.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 92 | 89 | 181
  Female | 12 | 11 | 23
  Unknown | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Unknown | 1 | 3 | 4
  Race: Black or African American | 10 | 9 | 19
  Race: White | 84 | 80 | 164
  Race: Other | 9 | 9 | 18
  Ethnicity: Unknown | 0 | 0 | 0
  Ethnicity: Not Hispanic or Latino | 98 | 95 | 193
  Ethnicity: Hispanic or Latino | 6 | 6 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 104 | 101 | 205
Education Completion [Count of Participants; unit: Participants]
  High school or less | 20 | 19 | 39
  Technical school | 5 | 4 | 9
  Some college | 52 | 51 | 103
  College degree or more | 27 | 27 | 54
Relationship Status [Count of Participants; unit: Participants]
  Married | 40 | 32 | 72
  Divorced/Separated | 36 | 38 | 74
  Widowed | 3 | 6 | 9
  Living together, not married | 10 | 5 | 15
  Never Married | 15 | 20 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinks Per Day as Assessed by Timeline Follow-Back (TLFB)
Description: Alcohol consumption is measured by Timeline Follow-Back (TLFB). The investigators will administer a 30-day TLFB for finer grained data on participant's self-reported drinking behaviors. The investigators will collect participant self-report data on number of drinks per day on days of drinking.
Time Frame: At 12-months post-randomization
Measure: Least Squares Mean (95% Confidence Interval); unit: Drinks per day
Arm/Group | Alcohol Peer-Mentor Intervention | Brief Advice
Number analyzed (Participants) | 104 | 101
Drinks per day | 0.91 [0.66 to 1.14] | 1.62 [1.18 to 2.02]

2. Primary Outcome: Number of Binge Drinking Days as Assessed by Timeline Follow-Back (TLFB)
Description: Alcohol consumption is measured by Timeline Follow-Back (TLFB). The investigators will administer a 30-day TLFB for finer grained data on participant's self-reported drinking behaviors. The investigators will collect participant self-report data on number of days when the participant demonstrates binge drinking (5+ drinks per day for men; 4+ drinks per day for women).
Time Frame: At 12-months post-randomization
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of Binge Drinking Days
Arm/Group | Alcohol Peer-Mentor Intervention | Brief Advice
Number analyzed (Participants) | 104 | 101
Number of Binge Drinking Days | 1.0 [0.2 to 1.8] | 3.7 [2.3 to 5.1]

3. Secondary Outcome: Frequency of Healthcare Utilization as Measured by Treatment Services Review (TSR, v6)
Description: The investigators will use the Treatment Services Review (TSR, v6) to measure the total number of healthcare visits across medical, mental health, and substance use care. The TSR, v6 is a semi-structured interview that gathers specific healthcare utilization information with adequate reliability and validity.
Time Frame: At 12-months post-randomization
Measure: Least Squares Mean (Standard Deviation); unit: number of clinic visits
Arm/Group | Alcohol Peer-Mentor Intervention | Brief Advice
Number analyzed (Participants) | 104 | 101
number of clinic visits
  Substance Use Disorder clinic visits | 3.0 (16.1) | 1.3 (5.7)
  Emergency Department visits | 1.2 (1.8) | 1.2 (1.5)

ADVERSE EVENTS:
Time Frame: 1 year, 3 months
Arm/Group | Alcohol Peer-Mentor Intervention | Brief Advice
All-Cause Mortality (participants affected / at risk) | 0/104 | 3/101
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/101
Other Adverse Events (participants affected / at risk) | 0/104 | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT03536546/Prot_SAP_000.pdf